CLINICAL TRIAL: NCT05626088
Title: Sociodemographic Characteristics, Vedolizumab Persistence and Outcomes in Inflammatory Bowel Disease Patients Participating in the Patient Support Program in Brazil
Brief Title: A Study in Adults With Inflammatory Bowel Disease (IBD) Receiving Vedolizumab in the Patient Support Program (PSP) in Brazil
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-4045; MACS-2022-042701 (Other: Takeda)
Record Dates: First submitted 2022-11-16; First posted 2022-11-23 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: Participants diagnosed with UC or CD with prescription of vedolizumab, and were included in the PSP program (which has started in 2016) before the study starts will be observed retrospectively in this study.
  Interventions: Other: No Intervention
- Prospective Cohort: Participants diagnosed with UC or CD with prescription of vedolizumab, and have participation in PSP after the study start will be observed prospectively in this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The primary reason of this study is to observe current and past treatment in adult participants receiving Vedolizumab, intravenous (IV) or subcutaneous (SC), for IBD in Brazil. There is no treatment involved in this study, this is only an observational review of past and ongoing treatment data relating to Vedolizumab treatment for IBD (including Ulcerative Colitis [UC] and Crohn's Disease [CD]).

DETAILED DESCRIPTION:
This is a non-interventional, observational study in participants with IBD participating in the PSP. This study will enroll approximately 2160 participants. The study is divided into two cohorts according to data collection:

* Retrospective Cohort
* Prospective Cohort

The retrospective cohort is for participants that were included in the PSP prior to study start. This retrospective cohort will have data of participants that are actively participating in the Program and only their retrospective data will be collected. The prospective cohort is for participants that are starting their participation in the PSP using their data from the consent date until the end of the study or until the discontinuation in the PSP or in the study.

Retrospective and prospective cohorts will be collected from the PSP database, which will be the only source of participants for this study.

This single country trial will be conducted in Brazil. The duration of this observational study will be approximately 26 months.

ELIGIBILITY:
Inclusion Criteria:

• Who participated or who will participate in the "Entre Nós" program and participant who consent to participate in the study.

Exclusion Criteria

• No exclusion of participants is expected in the present study and the quality of the data relies in participant reported outcomes for the "Entre Nós" program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with UC or CD with vedolizumab prescription, residing in Brazil and agree to participate in the program.
Sampling Method: Non-Probability Sample
Enrollment: 1006 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Vedolizumab Treatment Persistence for Conventional Therapy and Advanced Therapies | Up to approximately 9 years
  Treatment persistence will be defined as participants who did not discontinue treatment during follow-up. Advance therapies include biologics and tofacitinib.

SECONDARY OUTCOMES:
Number of Participants With Therapies Used Before Vedolizumab Treatment | Up to approximately 9 years
Number of Participants With Vedolizumab Treatment Scheme (Dose Escalation and De-escalation) for Conventional and Advanced Therapies | Up to approximately 9 years
  Advance therapies include biologics and tofacitinib.
Number of Participants With Comorbidities Associated or not With CD or UC | Up to approximately 9 years
Duration of Disease | Up to approximately 9 years
Percentage of Participants Diagnosed With UC or CD | Up to approximately 9 years
Percentage of Participants With Vedolizumab Drug Administration Route: Intravenous (IV) or Subcutaneous (SC) | Up to approximately 9 years
Number of Participants Based on Quality-of-life (QOL) as Assessed by Short Inflammatory Bowel Disease Questionnaire 10 (SIBDQ-10) in Prospective Cohort | At the index date (vedolizumab initiation), and at 14 and 52 weeks from index date
  The SIBDQ is a validated tool used by health care professionals for assessment of participant's inflammatory bowel disease. SIBDQ contains 10 (ten) questions, and each question is composed of the 7 (seven) levels of self-perception of feeling or mood, giving an absolute score ranging from 10 (poor health related QoL) to 70 (optimal health related QoL), higher scores mean better quality of life. Index date will be defined as the start of the vedolizumab treatment.
Percentage of Participants With Adverse Events (AEs) or Serious AEs During Vedolizumab use for UC and CD | Up to approximately 9 years
Number of Participants With Reason for Discontinuing the Vedolizumab Treatment for Conventional Therapy and Experiences Anti-TNF | Up to approximately 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Pesquisare Saúde S/S Ltda, Santo André, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/02e9c7fcf086437f?idFilter=%5B%22Vedolizumab-4045%22%5D